CLINICAL TRIAL: NCT05430152
Title: A Double Blind Randomized Trial of Low-dose Naltrexone for Post-COVID Fatigue Syndrome
Brief Title: Low-dose Naltrexone for Post-COVID Fatigue Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Luis Nacul (Other)
Collaborators: University of British Columbia (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Provincial Health Services Authority British Columbia (Other); Women's Health Research Institute of British Columbia (Other)
Responsible Party: Sponsor-Investigator, Luis Nacul, Clinical Associate Professor, University of British Columbia
Organization: University of British Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H21-02254
Record Dates: First submitted 2022-06-10; First posted 2022-06-24 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Post-Viral Fatigue Syndrome
Keywords: Post-COVID Fatigue Syndrome; Long-COVID; COVID-19; SARS-CoV-2
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Post-Acute COVID-19 Syndrome; COVID-19 | interventions — Naltrexone

STUDY DESIGN:
Intervention Model Description: Randomized parallel group double-blinded placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-Dose Naltrexone (Experimental): The Low-Dose Naltrexone (LDN) will be provided as a compounded capsule starting at a strength of 1mg/day of naltrexone and increasing up to a maximum of 4.5 mg/day. The compounding pharmacy will compound the needed doses in Capsugel® empty gelatin based capsules using Naltrexone Hydrochloride Tablets and CELLULOSE.
  Interventions: Drug: Low-Dose Naltrexone
- Placebo (Placebo Comparator): Matching placebo capsule will be created by compounding pharmacy to look exactly like the LDN doses. The compounding pharmacy will compound the placebo in Capsugel® empty gelatin based capsules using CELLULOSE.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Low-Dose Naltrexone — Study drug dosing schedule (LDN):
  * Week 1: 1 mg/day (1 mg cap)
  * Week 2: 2 mg/day (two 1 mg caps)
  * Week 3: 3 mg/day (three 1mg caps)
  * Weeks 4-6: 4.5 mg/day (three 1 mg caps, plus one 1.5 mg cap = 4.5 mg/day)
  * Weeks 7-16: 4.5 mg/day (one 4.5 mg cap) OR based on self-titration dosage (one 1mg, 2mg, or 3mg cap)
  Other Names: LDN
  Arms: Low-Dose Naltrexone
Other: Placebo — Study drug dosing schedule (Placebo; capsules made to match LDN doses):
  * Week 1: 1 mg/day (1 mg cap)
  * Week 2: 2 mg/day (two 1 mg caps)
  * Week 3: 3 mg/day (three 1mg caps)
  * Weeks 4-6: 4.5 mg/day (three 1 mg caps, plus one 1.5 mg cap = 4.5 mg/day)
  * Weeks 7-16: 4.5 mg/day (one 4.5 mg cap) OR based on self-titration dosage (one 1mg, 2mg, or 3mg cap)
  Arms: Placebo

SUMMARY:
This study aims to determine if low-dose naltrexone (LDN) reduces fatigue, improves related symptoms, and reduces inflammatory markers in peripheral blood in cases with Post-COVID-19 Fatigue Syndrome (PCFS) from COVID-19 (i.e. confirmed SARS-CoV-2 case). LDN refers to naltrexone given in doses of 1-4.5 mg. Overall, studies have found that LDN is safe and well-tolerated. It may help to reduce pain and inflammation and improve well-being and immune function.The trial will be conducted by the Complex Chronic Diseases Program (CCDP) at BC Women's Hospital and will demonstrate whether LDN could benefit a large number of people with PCFS.

DETAILED DESCRIPTION:
There is a growing number of individuals who do not recover to previous levels of health and function following an acute infection by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), but rather develop what has been referred to as 'Long-COVID'. Long-COVID is believed to be multi-causal, with a significant proportion of Long-COVID cases developing a clinical picture indistinguishable from myalgic encephalomyelitis/ chronic fatigue syndrome (ME/CFS) or post-viral fatigue syndrome (PVFS), which we will refer to as post-COVID-19 fatigue syndrome (PCFS). It is characterized by persistent disabling fatigue and other symptoms, such as nonrestorative sleep and post-exertional malaise. Diagnosis is clinical and based on symptom reports owing to the absence of diagnostic biomarkers. Viral and other infections are 25 times more likely to trigger ME/CFS than any other factors. This highlights the possibility of COVID-19 survivors having post-viral symptoms which progress to PCFS, either as the only sequelae or combined with other dysfunctions. Other Long-COVID symptom profiles in addition to PCFS include: a) post-intensive care syndrome; b) organ damage; and c) other debilitating symptoms related to mental health and other conditions.

There is no evidence-based treatment for PVFS, however, low-dose naltrexone (LDN), i.e. in doses up to 4.5 mg/day, has been used with some success in cases not related to COVID-19, due to its potential anti-inflammatory, analgesic properties and other mechanisms, targeting potential key mechanisms involved in the development of PVFS and the persistence of symptoms long-term.

Previous literature has demonstrated the safety and effectiveness of LDN in other chronic conditions, such as fibromyalgia (FM). The use of LDN as an off label treatment for fibromyalgia and myalgic encephalomyelitis has been used extensively within the BC Women's Hospital + Health Center's Complex Chronic Diseases Program (CCDP) to treat symptoms of pain and fatigue in these clinical populations. The experience of doctors in the CCDP in administering LDN as a medication for these related diseases follows international clinical experience with LDN and the recommended usage from clinical trials in fibromyalgia.

Naltrexone is an opiate antagonist approved by Health Canada for treatment for alcohol and opiate use disorders. It is used off label at low doses for conditions such as ME/CFS, fibromyalgia and Crohn's disease, with good safety profile and some evidence of benefit.

The impact the COVID-19 pandemic makes finding evidence for an effective and safe treatment for PCFS urgent. With currently no curative treatment for ME/CFS or PCFS, a larger number of people are predicted to be impacted by the long-term morbidity and disability associated with these conditions, with high costs to healthcare and social services.

The Double Blind Randomized Trial of Low-Dose Naltrexone for Post-COVID Fatigue Syndrome (PCFS) is a randomized parallel group double-blinded placebo-controlled trial of daily oral capsules of LDN or placebo for individuals 19-69 years old of both sexes for the treatment of PCFS. 160 participants will be treated with either LDN or placebo for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ages 19 to less than 70 years
2. Case of SARS-CoV-2 over 3 previously, confirmed by a positive test result or clinical confirmation by a physician
3. Meet the clinical diagnostic criteria for PCFS
4. Agree to maintain any other regular medications at current doses for the duration of the trial (except for essential need of new medication or dose change, as prescribed by a physician)
5. Agree to use effective contraception for the trial duration, as appropriate, if female.
6. The participant resides within the delivery area for the drug as determined by FedEx Clinical Trial Services

Exclusion Criteria:

1. Pregnant, planning to become pregnant, or breastfeeding
2. Opioid medications:

   * Any use within last 15 days, as reported by the patient
   * During the trial
3. A positive urine test for opioids (only for the first 16 participants)
4. History of alcohol, opioid or other substance misuse
5. Participation in another interventional clinical trial in the last 30 days or planned during the trial period
6. Confirmed ME/CFS or FM existing prior to SARS-CoV-2 infection
7. Allergy to naltrexone or medication components
8. Acute hepatitis, liver failure, or severe kidney failure.
9. Current or recent use of naltrexone in the last 30 days
10. The participant is not an ideal candidate for the study, in the opinion of the investigator, for any other reason (ie. personal or logistic, medication, condition, etc.) that could impact the participant's safety or the results of the study.

Opioid Washout Period:

Potential participants who are currently taking opioid medications who wish to enrol the study will be instructed they can stop taking opioid medications for 15 days before continuing the screening process. They will be instructed that they should speak with their family doctor before stopping any prescribed medications.

Positive Urine Test for Opioids:

As regular use of opioid medications is an exclusion criterion, we will do a quality control check with the first 16 participants to test for the presence of opioids in their urine. Any participants with a positive test, will be excluded from the study, and such finding will be discussed at the Trial Steering Committee or DSMB for potential trial modification.

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-08-16 (Estimated); Study Completion 2025-08-16 (Estimated)

PRIMARY OUTCOMES:
Fatigue Intensity | 16 weeks
  Change in the Fatigue Severity Scale (FSS) total score by 4.7 points or over

SECONDARY OUTCOMES:
Pain Severity | 16 weeks
  Change in Pain Visual Analogue Scale (VAS) 0-10 score
Symptom Severity | 16 weeks
  Change in Patient Phenotyping Questionnaire Short Form (PQSymp-12) score
Activity Levels | 16 weeks
  Changes in average number of steps over 7 days
Self-reported Quality of Life | 16 weeks
  Change in EuroQol-5 Dimension 5-level (EQ-5D-5L) total score

OTHER OUTCOMES:
Exploratory outcome: Changes in inflammatory marker values in peripheral blood | 16 weeks
  Changes in Interleukin 6 (IL-6), Interferon gamma (IFNγ), C-reactive protein (hsCRP), & cytokine profile (Human High Sensitivity T-Cell 14-plex Discovery Assay® Array) values
Exploratory outcome: Disease Severity | 16 weeks
  Change in Creatine kinase (CK) plasma concentration
Exploratory outcome: Reverse triiodothyronine (rT3) profile (as an indirect marker of disease severity) | 16 weeks
  Change in concentration of Reverse triiodothyronine (rT3) (in conjunction Thyroid stimulating hormone (TSH), Free Triiodothyronine (free T3) & Free Thyroxine (free T4))
Exploratory outcome: Visual Analogue Scale (VAS) Fatigue Score | 16 weeks
  Change in the fatigue Visual Analogue Scale (VAS) 0-10 score
Exploratory outcome: Prevalence markers of Postural Orthostatic Tachycardia Syndrome (POTS) or Postural Hypotension | 16 weeks
  Change in the prevalence of POTS or postural hypotension symptoms based on serial blood pressure and heart rate measurement
Exploratory outcome: Sleep SQ-2 | 16 weeks
  Changes in the Sleep Questionnaire (SQ-2)
Exploratory outcome: Sleep-VAS | 16 weeks
  Changes in the self-reported sleep Visual Analogue Scale (VAS)
Exploratory outcome: Depression | 16 weeks
  Changes in the Patient Health Questionnaire (PHQ-9) Score
Exploratory outcome: Anxiety | 16 weeks
  Changes in the Generalized Anxiety Disorder (GAD-7) Score
Exploratory outcome: Self-reported Health | 16 weeks
  Changes in the self-reported Visual Analogue Scale (VAS) health scale (EQ-5D-5L)
Exploratory outcome: Improves low AM blood cortisol | 16 weeks
  Changes in concentration of AM blood cortisol values
Exploratory outcome: Improves Adrenocorticotropic hormone (ACTH) | 16 weeks
  Changes in concentration of ACTH hormone values
Exploratory outcome: Improves Functional Status | 16 weeks
  Changes in Post-COVID-19 Functional Status Scale
Clinical Endurance/ Hand Grip Strength Parameters | 16 weeks
  Changes in maximum hand grip strength over 3 attempts
Clinical Endurance/ Sit and Stand Strength Parameters | 16 weeks
  Changes in sit and stand test in 30 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Luis Nacul, MD, PhD, Principal Investigator — WHRI / University of British Columbia
Locations (1):
- Women's Health Research Institute, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
At the time of publication, the study data may be deposited on a publicly accessible location.
Supporting Information: Study Protocol
Time Frame: Protocol has been shared in peer-reviewed paper
Access Criteria: open access
URL: https://bmjopen.bmj.com/content/14/5/e085272

REFERENCES:
- [Derived] Naik H, Cooke E, Boulter T, Dyer R, Bone JN, Tsai M, Cristobal J, McKay RJ, Song X, Nacul L. Low-dose naltrexone for post-COVID fatigue syndrome: a study protocol for a double-blind, randomised trial in British Columbia. BMJ Open. 2024 May 13;14(5):e085272. doi: 10.1136/bmjopen-2024-085272. PMID 38740499